CLINICAL TRIAL: NCT01704404
Title: A Phase 2 Study of the Pharmacodynamics, Safety and Tolerability, and Pharmacokinetics of Multiple Doses of TD-4208 for 7 Days in Subjects Diagnosed With Chronic Obstructive Pulmonary Disease
Brief Title: 7 Days of TD-4208 in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0091
Record Dates: First submitted 2012-10-04; First posted 2012-10-11 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: COPD
Keywords: Long acting muscarinic antagonist; Chronic Bronchitis; Emphysema; Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — revefenacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Dose 1 TD-4208 (Experimental): 22 µg
  Interventions: Drug: TD-4208
- Dose 2 TD-4208 (Experimental): 44 µg
  Interventions: Drug: TD-4208
- Dose 3 TD-4208 (Experimental): 88 µg
  Interventions: Drug: TD-4208
- Dose 4 TD-4208 (Experimental): 175 µg
  Interventions: Drug: TD-4208
- Dose 5 TD-4208 (Experimental): 350 µg
  Interventions: Drug: TD-4208
- Dose 6 TD-4208 (Experimental): 700 µg
  Interventions: Drug: TD-4208
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-4208
  Other Names: revefenacin
  Arms: Dose 1 TD-4208; Dose 2 TD-4208; Dose 3 TD-4208; Dose 4 TD-4208; Dose 5 TD-4208; Dose 6 TD-4208
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will characterize the dose response of TD-4208 after 7 days of dosing in subjects with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female between the ages of 40 and 75 years (inclusive, at randomization).
2. Subject:

   * Has an FEV1/FVC (forced expiratory volume in 1 second/forced vital capacity) <0.7 at screening; and
   * Has a post-bronchodilator FEV1 at screening of between 30% and 80% (inclusive) of the predicted normal value.
3. Subject demonstrates at screening at least a 120 mL increase in FEV1 within 1 hour of receiving 500 µg of ipratropium bromide from a PARI LC Sprint® nebulizer.
4. Females of non-childbearing potential. All male subjects must agree to use a highly effective method of birth control with partners of childbearing potential during the study and for 1 month after completion of study dosing.
5. Subject (or care giver) is able to properly prepare and administer study medication.
6. Subject is willing and able to give written informed consent to participate.

Exclusion Criteria:

1. Subject has had a COPD exacerbation or lung infection within 6 weeks before randomization.
2. Subject has had an initiation of treatment, or a change in dose, of an inhaled or oral corticosteroid, or long-acting beta2 agonist (LABA), or long-acting muscarinic antagonist (LAMA) within 4 weeks before the qualifying ipratropium bromide response test.
3. Subject is taking daily maintenance inhaled/systemic corticosteroids (>1000 μg of fluticasone propionate equivalent or ≥10 mg prednisone).
4. Subject has an uncontrolled hematologic, immunologic, renal, neurologic, hepatic, endocrine, or other disease or condition based on information gathered from the medical history, physical examination, or laboratory findings that might place the subject at undue risk or potentially compromise the results or interpretation of the study.
5. Subject has a history of significant cerebrovascular disease, coronary artery disease, or cardiac arrhythmias. Subject has a history (or family history) of congenital prolonged QTc (corrected QT interval) syndrome or has an abnormal clinically significant electrocardiogram (ECG) at screening, including QTcB (QT interval corrected for heart rate using Bazett's formula) value >450 msec (males) or >470 msec (females); or shows evidence of clinically significant rhythm abnormality.
6. Subject has a known hypersensitivity to TD-4208 or similar drug class.
7. Subject has a history of alcoholism or drug abuse within 2 years prior to screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- P3 Research Ltd, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo A, Borin MT, Bourdet DL. Population Pharmacokinetics of Revefenacin in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2021 Mar;60(3):391-401. doi: 10.1007/s40262-020-00938-3. PMID 33124005
- [Derived] Quinn D, Barnes CN, Yates W, Bourdet DL, Moran EJ, Potgieter P, Nicholls A, Haumann B, Singh D. Pharmacodynamics, pharmacokinetics and safety of revefenacin (TD-4208), a long-acting muscarinic antagonist, in patients with chronic obstructive pulmonary disease (COPD): Results of two randomized, double-blind, phase 2 studies. Pulm Pharmacol Ther. 2018 Feb;48:71-79. doi: 10.1016/j.pupt.2017.10.003. Epub 2017 Oct 4. PMID 28987804

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1: Placebo, 44 µg, 88 µg, 350 µg, 700 µg
- Treatment 2: Placebo, 22 µg, 88 µg, 350 µg, 700 µg
- Treatment 3: Placebo, 22 µg, 88 µg, 175 µg, 700 µg
- Treatment 4: 22 µg, 44 µg, 175 µg, 700 µg
- Treatment 5: 22 µg, 44 µg, 175 µg, 350 µg
- Treatment 6: Placebo, 44 µg, 88 µg, 175 µg, 350 µg
Period: Overall Study
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment 6
Started | 11 | 10 | 10 | 11 | 11 | 9
Completed | 10 | 9 | 9 | 8 | 10 | 9
Not Completed | 1 | 1 | 1 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All subjects received Placebo and 4 of 6 TD-4208 dose levels:
  TD-4208 - 22 µg TD-4208 - 44 µg TD-4208 - 88 µg TD-4208 - 175 µg TD-4208 - 350 µg TD-4208 - 700 µg
Arm/Group | Entire Study Population
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: year] | 64.2 (6.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 7 in Trough FEV1 (Forced Expiratory Volume in 1 Second)
Time Frame: From baseline to day 7
Measure: Mean (Standard Error); unit: FEV1 (mL)
Groups:
- Dose 1 TD-4208: 22 µg
  TD-4208
- Dose 2 TD-4208: 44 µg
  TD-4208
- Dose 3 TD-4208: 88 µg
  TD-4208
- Dose 4 TD-4208: 175 µg
  TD-4208
- Dose 5 TD-4208: 350 µg
  TD-4208
- Dose 6 TD-4208: 700 µg
  TD-4208
Arm/Group | Dose 1 TD-4208 | Dose 2 TD-4208 | Dose 3 TD-4208 | Dose 4 TD-4208 | Dose 5 TD-4208 | Dose 6 TD-4208 | Placebo
Number analyzed (Participants) | 40 | 39 | 39 | 39 | 39 | 40 | 59
FEV1 (mL) | 91.2 (19.21) | 92.8 (20.25) | 113.1 (19.55) | 151.9 (19.99) | 132.2 (19.02) | 119.4 (19.54) | 37.8 (16.93)

2. Other Pre Specified Outcome: Cmax
Description: Day 1: 15 minutes pre-dose, post-dose at 15 and 30 minutes, 1, 2, 3, 4, and 6 hours.
  Day 7: 15 minutes pre-dose, post-dose at 15 and 30 minutes, 1, 2, 3, 4, 6, 8, 12 and 24 hours.
Time Frame: From baseline to day 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose 1 TD-4208 | Dose 2 TD-4208 | Dose 3 TD-4208 | Dose 4 TD-4208 | Dose 5 TD-4208 | Dose 6 TD-4208
Number analyzed (Participants) | 37 | 36 | 35 | 35 | 40 | 35
ng/mL | .0125 (.00627) | .0224 (.00864) | .0526 (.0214) | .114 (.0488) | .243 (.104) | .577 (.261)

3. Other Pre Specified Outcome: Tmax
Description: as for outcome 2
Time Frame: From baseline to day 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose 1 TD-4208 | Dose 2 TD-4208 | Dose 3 TD-4208 | Dose 4 TD-4208 | Dose 5 TD-4208 | Dose 6 TD-4208
Number analyzed (Participants) | 37 | 36 | 35 | 35 | 40 | 35
hours | .233 (.217) | .233 (0.200) | 0.233 (0.200) | 0.233 (0.200) | 0.233 (0.217) | 0.233 (0.200)

4. Other Pre Specified Outcome: Plasma Half-life
Description: as for outcome 2
Time Frame: From baseline to day 7
Population: The number of subjects reported for plasma half lives are based on the actual evaluable PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose 1 TD-4208 | Dose 2 TD-4208 | Dose 3 TD-4208 | Dose 4 TD-4208 | Dose 5 TD-4208 | Dose 6 TD-4208
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 31 | 26
hours |  |  |  |  | 25.1 (7.89) | 23.0 (7.05)

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: The Participant Flow shows the # of subjs in each of the 6 treatment sequences (each sequence has 4 treatments; 4/6 study drug doses and placebo) as instructed by CTgov for complex crossover designs. The Number of Participants at Risk, instead, shows the # of subjs exposed to each of the 6 doses of study drug and placebo. Also, some subjs did not complete all of the doses in their treatment sequence. The # of subjs in each sequence is not related to the # of subjs in each dose level therefore.
Arm/Group | Dose 1 TD-4208 | Dose 2 TD-4208 | Dose 3 TD-4208 | Dose 4 TD-4208 | Dose 5 TD-4208 | Dose 6 TD-4208 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/42 | 0/42 | 0/40 | 0/41 | 0/41 | 0/42 | 1/62
Other Adverse Events (participants affected / at risk) | 14/41 | 12/39 | 12/40 | 13/37 | 8/41 | 9/37 | 16/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 TD-4208 (N=42) | Dose 2 TD-4208 (N=42) | Dose 3 TD-4208 (N=40) | Dose 4 TD-4208 (N=41) | Dose 5 TD-4208 (N=41) | Dose 6 TD-4208 (N=42) | Placebo (N=62)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 TD-4208 (N=41) | Dose 2 TD-4208 (N=39) | Dose 3 TD-4208 (N=40) | Dose 4 TD-4208 (N=37) | Dose 5 TD-4208 (N=41) | Dose 6 TD-4208 (N=37) | Placebo (N=61)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 5 (5) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.